CLINICAL TRIAL: NCT00442975
Title: A Phase IV, Single Group Study to Evaluate the Immune Response to Licensed Seasonal Influenza Vaccine and Relationship of This to Cytomegalovirus-associated Immunosenescence in UK Older Adults Aged 50-80 Years
Brief Title: Response of Older Adults to Influenza Vaccination With Regard to Cytomegalovirus (CMV) Status
Acronym: CMVflu
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Public Health England (Other Government)
Collaborators: Royal Free and University College Medical School (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: CMVfluvaccinees; EudraCT No: 2006-006563-23
Record Dates: First submitted 2007-03-02; First posted 2007-03-05 (Estimated); Last update posted 2018-08-29 (Actual); Status verified 2008-02

CONDITIONS: Influenza
Keywords: Influenza Vaccine; CMV
MeSH Terms: conditions — Influenza, Human | interventions — fluarix

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Biological: Fluarix

SUMMARY:
The study is being undertaken to evaluate responses to seasonal influenza vaccine in older adults with respect to their CMV status. CMV is cytomegalovirus and is an organism that infects many people, but does not usually cause disease in the individual unless they are immunocompromised i.e. their immune system is not working well such as in the case of HIV infection. CMV is believed to have infected up to 80% of individuals in the age group we will be looking at in our study and we are interested in whether this infection affects their responses to vaccination.

DETAILED DESCRIPTION:
Human cytomegalovirus (HCMV) is an important pathogen or disease-causing virus, which can result in disease in the unborn child as well as in individuals whose immune systems are not working properly such as those with HIV or who are receiving some treatments for cancer, where the body's ability to fight infection is not as good as in healthy people. HCMV infects the majority of the population, yet rarely causes overt disease which would limit the capacity of the host to transmit HCMV to others. This virus is thought to be millions of years old and because of this we think that it has evolved over time to become very efficient at evading the immune system. This means it has become very efficient at moving through the human population and resulting in humans devoting more immunological resources to controlling this virus than to any other. Recent studies have reported that the immune system does work less efficiently in older people, especially in elderly patients with CMV antibodies compared to age matched controls who did not have CMV antibodies.

It is well recognized that responses to vaccination are generally lower in older populations compared to children, so they may be thought to be immunologically in a suboptimal position. It is proposed that this may be as a result of diversion of key factors in the immune system to address CMV infection, the incidence of which increases with age. This study will allow assessment of responses to licensed seasonal influenza vaccine with respect to age and CMV status and will provide baseline information as a proof of principle on which a larger study will be designed.

ELIGIBILITY:
Inclusion Criteria:

* No contraindications to vaccination as specified in the "Green Book" - Immunisation Against Infectious Disease, HMSO.
* Written informed consent obtained
* Subject aged no less than 50 years 0 days and no older than 79 years and 364 days at enrollment.

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2007-03; Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
Response to influenza vaccination (HI)

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Miller, MBBS FRCPath, Principal Investigator — Public Health England
Locations (1):
- Hertfordshire Primary Care Trust, Stevenage, United Kingdom